CLINICAL TRIAL: NCT07093541
Title: An Open Label Expanded Access Program Intended to Provide Treatment With Ecopipam (EBS-101) to Children, Adolescents, and Adults in the U.S. With Tourette's Disorder
Brief Title: Expanded Access Program for Treatment With Ecopipam for Tourette's Disorder
Acronym: EBS-101-TD-392
Status: Available | Type: Expanded Access
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EBS-101-TD-392
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Tourettes Disorder; Tourette Disorder
Keywords: Tourettes Syndrome; Ecopipam Tourette Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: ecopipam HCl ~2mg/kg/day — Daily oral tablet taken every evening before bedtime.
  Other Names: EBS-101

SUMMARY:
The goal of this expanded access study is to learn about the long-term effects of Ecopipam in participants with Tourette's Disorder (TD). The main question it aims to answer is:

* Is ecopipam safe and well-tolerated in participants equal and over the age of 6 to 50 with TD?
* Assess quality of life measures and to provide access to ecopipam while NDA is being prepared and submitted for review for marketing approval

Eligible participants with TD will take ecopipam with guidance from their treating physician. In addition to the standard of care from the treating physician, treatment with ecopipam will continue until ecopipam becomes commercially available in the United States or the program is terminated.

While in the EAP program, participants will be asked regarding how safe and tolerable ecopipam is to the participant. Several questionnaires will be collected regarding participants experiences while taking ecopipam during monthly visits for the first year and every three months thereafter until the conclusion of the study.

DETAILED DESCRIPTION:
The main purpose of this study is to further study the safety and tolerability of ecopipam in children, adolescents, and adults with Tourette's Disorder (TD).

The secondary objectives of this program are to assess patient-reported outcome measures including quality of life (QOL) and to provide access to ecopipam while a U.S. New Drug Application (NDA) is being prepared and submitted for review for marketing approval in the U.S.

This is an open label expanded access program for ecopipam (EBS-101) intended to collect safety information and physician-administered psychiatric scales and patient-reported outcomes in children, adolescents, and adults in the U.S. with TD who are unable to take currently approved medications for TD (aripiprazole, haloperidol, or pimozide) or any other D2 receptor antagonists (D2rA) due to treatment failure, intolerability, safety or lack of access.

At the Screening visit, participants will provide informed consent [adult participants or children/adolescent Legally Acceptable Representative (LAR)] and assent (children/adolescents) and be assessed against the inclusion/exclusion criteria for participation in the study. Demographic information, disease comorbidities, and concomitant medications will be documented, vital signs and a physical examination will be performed, blood and urine samples will be collected for safety laboratories, an electrocardiogram (ECG) will be performed, lifetime history for suicidality will be assessed using the Columbia Suicidality Severity Rating Scale (C-SSRS), and age group validated scales to assess anxiety and depression will be performed. The participant and in the case of pediatric participants their LAR will also be asked to complete scales to assess the severity of their disease and quality of life.

Based on satisfying Screening visit criteria, participants will receive a telephone call to confirm Enrollment (Day 1). Visit dates will be defined from date of first dose. Once Enrollment is confirmed, eligible participants will be registered with a specialty pharmacy who will dispense ecopipam. Participants will be gradually titrated over a period of 2-4 weeks depending on their weight to achieve a target steady-state dose of 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam HCl).

Following the Enrollment call, there will be a telemedicine assessment in approximately 2 weeks to assess adverse events (AEs) and participant tolerance to ecopipam. Participants will return to the clinic at monthly intervals for safety and efficacy assessments for the first year of treatment and every 3 months thereafter until study termination as outlined in the Schedule of Assessments (Table 5).

Participants will also be contacted 30 days after the last dose of study drug to determine any additional AEs or concomitant medications, to administer the C-SSRS and to confirm compliance with taper down medication and study drug return.

ELIGIBILITY:
Participants must fulfill all of the following inclusion criteria to be eligible for participation in the Study:

1. Age 6 to 50 years old inclusive at the time of informed consent/assent.
2. Participant must sign/date the most current Informed Consent Form (ICF). For minor participants the LAR must/sign date the most current consent and the participant must sign/date the most current age-appropriate assent.
3. In the opinion of the principal investigator (PI), the participant or in the case of a minor their LAR is capable of understanding and complying with protocol and program requirements, oral drug administration and care instructions.
4. Weight ≥18 kg (39.6 lbs.).
5. In the opinion of the PI, the participant meets diagnostic criteria for Tourette's Syndrome (TS) per Diagnostic and Statistical manual for Mental Disorders - 5th Edition (DSM-5-TR diagnostic criteria for TD).
6. The participant must have been treated with an FDA-approved treatment for TD (aripiprazole, haloperidol, or pimozide) or any other D2r antagonist (D2rA) and have experienced treatment failure, tolerability or safety issues as per LAR, participant or prescribing clinician or not have access to any of these approved medications.
7. Females of child-bearing potential must have a negative urine pregnancy test at Screening.
8. Females of child-bearing potential who are sexually active or become sexually active must be using double barrier method (condom and IUD, condom and spermicide, etc.) in addition to any oral contraceptive they may be using and agree to continue use of double barrier contraception for the duration of their participation in the study and for 30 days after their last dose of study drug. Females of non-childbearing potential are exempt from this criterion.

   Non-Childbearing potential is defined by:
   1. Post menopausal defined as >= 2 years amenorrheic, or,
   2. Bilateral salpingo-oopherectomy, or
   3. Hysterectomy, or
   4. Pre-menarche
9. Sexually active male participants must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.
10. Male participants must agree to not donate sperm and female participants not to donate eggs for at least 30 days after the last dose of study drug.

Diagnosis and Main Criteria for Inclusion:

Inclusion Criteria

Participants must fulfill all of the following inclusion criteria to be eligible for participation in the Study:

1. Age 6 to 50 years old inclusive at the time of informed consent/assent.
2. Participant must sign/date the most current Informed Consent Form (ICF). For minor participants the LAR must/sign date the most current consent and the participant must sign/date the most current age-appropriate assent.
3. In the opinion of the principal investigator (PI), the participant or in the case of a minor their LAR is capable of understanding and complying with protocol and program requirements, oral drug administration and care instructions.
4. Weight ≥18 kg (39.6 lbs.).
5. In the opinion of the PI, the participant meets diagnostic criteria for Tourette's Syndrome (TS) per Diagnostic and Statistical manual for Mental Disorders - 5th Edition (DSM-5-TR diagnostic criteria for TD).
6. The participant must have been treated with an FDA-approved treatment for TD (aripiprazole, haloperidol, or pimozide) or any other D2r antagonist (D2rA) and have experienced treatment failure, tolerability or safety issues as per LAR, participant or prescribing clinician or not have access to any of these approved medications.
7. Females of child-bearing potential must have a negative urine pregnancy test at Screening.
8. Females of child-bearing potential who are sexually active or become sexually active must be using double barrier method (condom and IUD, condom and spermicide, etc.) in addition to any oral contraceptive they may be using and agree to continue use of double barrier contraception for the duration of their participation in the study and for 30 days after their last dose of study drug. Females of non-childbearing potential are exempt from this criterion.

   Non-Childbearing potential is defined by:
   1. Post menopausal defined as >= 2 years amenorrheic, or,
   2. Bilateral salpingo-oopherectomy, or
   3. Hysterectomy, or
   4. Pre-menarche
9. Sexually active male participants must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.
10. Male participants must agree to not donate sperm and female participants not to donate eggs for at least 30 days after the last dose of study drug.

Participants cannot be enrolled in the study if they meet any of the following criteria.

1. Clinically meaningful abnormalities on laboratory tests at Screening as determined by the PI.
2. Specific laboratory findings at enrollment

   1. T. Bili >= 2.5 x ULN for age (Participants with a history of Gilbert's Disorder must have prior documentation of the disorder.)
   2. ALT >= 2.5 x ULN for age
   3. AST >= 2.5 x ULN for age
   4. Positive urine drug screen for cocaine, amphetamine, benzodiazepines, barbiturates, phencyclidine (PCP), or opiates at Screening, except those receiving stable, prescribed treatment for attention deficit/hyperactivity disorder (ADHD) or a positive for benzodiazepine prescribed (either routine or as needed) for any anxiety disorder or anxiety associated with a depressive disorder
   5. Severe renal impairment or end stage renal disease as defined by eGFR < 60 ml/min/1.73m2
3. Any of the following cardiovascular:

   1. ECG with a QTcF > 450 for males or > 470 for females at screening.
   2. A history or finding on the screening ECG of any significant arrhythmia in the opinion of the principal investigator
   3. A known family history of QT prolongation syndrome with sudden death
   4. Current or anticipated need for medications known to prolong the QT interval
4. A lifetime history of any of the following disorders:

   1. Myocardial Infarction
   2. Cancer (excluding Basal Cell Carcinoma or Cervical Cancer in situ)
   3. Seizure Disorder (except febrile seizure)
   4. Neuroleptic Malignant Syndrome
   5. Tardive Dyskinesia
   6. Parkinson's Disorder
   7. Dementia
   8. Essential Tremor
   9. Substance Use Disorders (as defined by DSM-5-TR) in the past 6 months prior to screening. (Excluding nicotine and/or caffeine)
   10. Any general medical disorders OR psychiatric disorder that are not under good control in the opinion of the PI OR require treatment with any prohibited medication.
5. All prescription or over-the-counter drug (e.g., St. Johns Wort) that are strong and moderate inhibitors or inducers of CYP3A4; drugs that are substrates of CYP2D6; or drugs that are substrates of MATE-2K transporters (e.g., metformin).
6. At significant risk of attempting suicide in the opinion of the PI or any one of the following:

   1. A history of a suicide attempt OR behavior in the past one year prior to Screening.
   2. A lifetime history of 2 or more suicide attempts OR behaviors.
   3. A history of non-suicidal self-injurious behavior in the past 2 years prior to Screening.
   4. A history of suicide ideation OR thoughts in the past 6 months prior to Screening.
7. Female participants who are currently pregnant or lactating or planning to become pregnant during the study.
8. A history of hypersensitivity or allergic reaction to ecopipam or any inactive ingredient of the formulation.
9. Participants unable to swallow tablets.
10. Any participant who in the opinion of the PI or the Sponsor is not a suitable candidate for the program.

Ages: 6 Years to 50 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Atkinson, MD, Study Director — Emalex Biosciences